CLINICAL TRIAL: NCT03639649
Title: STHLM3 - Prostate Cancer Diagnostic Trial
Acronym: STHLM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Henrik Grönberg, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Karolinska1
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STHLM3 (Experimental)
  Interventions: Diagnostic Test: STHLM3
- PSA (Active Comparator)
  Interventions: Diagnostic Test: STHLM3

INTERVENTIONS:
Diagnostic Test: STHLM3

SUMMARY:
STHLM3 is a paired diagnostic trial aiming to assess whether a panel of biomarkers for prostate cancer can substantially reduce the proportion of men referred to biopsy whilst maintaining sensitivity for aggressive prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Age 50-69
* Residential address in Stockholm County

Exclusion Criteria:

* Previous Prostate Cancer Diagnosis
* Not able to comprehend inform consent material

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58818 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of biopsies | Recorded directly after biopsy

SECONDARY OUTCOMES:
Number of Gleason Score ≥ 7 | Recorded directly after biopsy
Number of Gleason Score 6 | Recorded directly after biopsy
Number of benign | Recorded directly after biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No